CLINICAL TRIAL: NCT00806663
Title: A Prospective Angiogenic Imaging Study With DCE-MRI and DCE-USI in Patients With Colorectal Cancer and Liver Metastases Receiving Sunitinib in Addition to 5-FU, Folinic Acid and Irinotecan (FOLFIRI) as 1st Line Therapy
Brief Title: FOLFIRI and Sunitinib in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Society for Anticancer Drug Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-II-005 /2008-001515-37
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Colorectal Cancer; Liver Metastases
Keywords: mCRC; colorectal cancer; FOLFIRI; sunitinib; DCE-MRI; DCE-USI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Arm (Experimental): Sutent sunitinib 37 mg once daily (4 weeks on/2 weeks off)
  Interventions: Drug: sunitinib added to FOLFIRI

INTERVENTIONS:
Drug: sunitinib added to FOLFIRI — sunitinib 37 mg once daily (4 weeks on/2 weeks off)
  Other Names: Sutent

SUMMARY:
This is an open label single arm prospective multicenter Phase II study in around 20 patients. The primary objective of this study is to evaluate whether the addition of sunitinib to FOLFIRI results in a significant reduction of tumor vessel permeability (TVP) and blood flow (BF) measured by DCE-MRI and DCE-USI, measured on liver metastases.

Secondary objectives are antitumor response, time to progression (TTP), effect on pharmacokinetics of sunitinib and biomarkers (VEGF und soluble VEGF-receptor) and drug/treatment safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females: over 18 years of age.
* Patients with histologically or cytologically confirmed colorectal cancer who will receive their first palliative treatment.
* Patients who have at least one measurable hepatic lesion of 2 cm or more according to RECIST criteria.
* ECOG 0 or 1.
* Signed written informed consent.
* White blood cell count (WBC)>= 4x10^9/L with neutrophils >= 1.5 x 10*9/L, platelet count >= 100x10*9/L, hemoglobin >= 5.6 mmol/L (10 g/dL).
* Total bilirubin =< 2 x upper limit of normal.
* AST and ALT =< 2.5 x upper limit of normal, or =< 5 x upper limit of normal in case of liver metastases.
* Serum creatinine =< 1.5 x upper limit of normal or creatinine clearance > 60 ml/min
* Normal ECG without QT prolongation.

Exclusion Criteria:

* Resectable liver metastasis.
* Adjuvant therapy with FOLFOX or 5-FU / Capecitabine =< 6 months prior to treatment on study or any previous palliative chemotherapy..
* Any contraindication for FOLFIRI chemotherapy regimen.
* Any investigational drug within the 30 days before inclusion.
* Prior use of sunitinib or other multitarget tyrosine kinase inhibitors or VEGF pathway directed treatments like bevacizumab.
* Known or suspected allergy or hypersensitivity reaction to any of the components of study treatments.
* Pregnancy (absence to be confirmed by beta-hCG test) or lactation period
* Men or women of child-bearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial
* Clinically symptomatic brain or meningeal metastasis. (known or suspected)
* Cardiac arrhythmias requiring anti-arhythmics (excluding beta blockers or digoxin).
* History of any of the following cardiac events within the past 6 months:

  * myocardial infarction (including severe/ unstable angina),
  * coronary/peripheral artery bypass graft,
  * congestive heart failure (CHF),
  * cerebrovascular accident,
  * transient ischemic attack pulmonary embolism.
* History of clinically significant bleeding within the past 6 months, including gross hemoptysis or haematuria, or underlying coagulopathy.
* History of peptic ulcer disease, deep vein thrombosis, or other significant thrombo-embolic event within the past 6 months.
* Uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 90 mm Hg despite the use of >= 3 anti-hypertensive drugs.
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease or chronic diarrhea.
* Previous malignancy (other than colorectal cancer) in the last 5 years except basal cell cancer of the skin, pre-invasive cancer of the cervix or superficial bladder tumor [Ta, Tis and T1].
* History of organ allograft
* Treatment with potent CYP3A4 inhibitor within 7 days of sunitinib/placebo dosing or with potent CYP3A4 inducer within 12 days of sunitinib/placebo dosing.
* Prior full field radiotherapy =< 4 weeks, or limited field radiotherapy, =< to 2 weeks prior to study enrollment; or previous radiation treatment >30% of the bone marrow.
* Major surgical procedure, open biopsy or significant traumatic injury within 4 weeks before starting treatment; anticipation of need for major surgical procedure (e.g. impending bowel obstruction) during the course of the study.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment, unless affected area has been removed surgically.
* Significant disease which, in the investigator's opinion would exclude the patient from the study.
* Patients with seizure and epileptic disorder or other conditions requiring medication such as phenytoin, carbamazepin, phenobarbital.
* Patients requiring long-term cortisone therapy.
* Patients requiring oral anticoagulation treatment (marcoumar).
* Known alcohol or drug abuse.
* Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
reduction of tumor vessel permeability (TVP) and blood flow (BF) measured by DCE-MRI and DCE-USI, measured on liver metastases. | 12 weeks

SECONDARY OUTCOMES:
Antitumour response | 9 months
Time to progression (TTP) | 9 months
pharmacokinetics | 12 weeks
drug treatment safety | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mross, MD, Study Chair — Klinik für Tumorbiologie
Locations (4):
- Germany (4):
  - Innere Univ.-Klinik u. Poliklinik Tumorforschung, Essen
  - Klinik für Tumorbiologie, Freiburg im Breisgau
  - Medizinische Universitätsklinik der Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau
  - Marienhospital, Herne